CLINICAL TRIAL: NCT06914297
Title: Immune Checkpoint Inhibitors Combined With Progestins for Fertility-sparing Treatment in Patients With MMRd Endometrial Cancer: a Multicenter Single-arm Prospective Clinical Trial
Brief Title: TQB2450 Plus Progestin for Fertility-sparing Treatment in MMRd EC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Vice President, Tenth People's Hospital of Tongji University, Shanghai, China, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FST-dMMR-ICIs
Record Dates: First submitted 2025-03-20; First posted 2025-04-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; Immune checkpoint inhibitor; fertility-sparing treatment; dMMR
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Progestins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICI plus P (Experimental): Initial hysteroscopic lesion resection and endometrial pathological evaluation were performed in patients who met the nanoparticle criteria, and drug therapy was initiated within one week: TQB2450 (1200 mg q3w ivgtt) + meprogesterone acetate (MA, 160 mg qdpo)/medroxyprogesterone acetate (MPA, 500 mg qdpo). Comprehensive/individualized hysteroscopic evaluation was performed at 12 weeks of treatment. According to the endometrial pathological results, radical surgery was recommended if the disease progressed (PD); if complete response/partial response (PR)/stable disease (SD) was achieved, the above regimen was continued with TQB2450 + MA/MPA. After 12 weeks of treatment, hysteroscopic comprehensive/individualized evaluation was performed again. According to the endometrial pathological results, if PR/SD/PD, radical surgical treatment was recommended. After treatment reached CR, the above regimen was continued to TQB2450 + MA/MPA consolidation treatment for 12 weeks.
  Interventions: Drug: TQB2450 injection + oral progestin

INTERVENTIONS:
Drug: TQB2450 injection + oral progestin — TQB2450 (1200 mg q3w ivgtt) + megestrol acetate (MA, 160 mg qd po)/megestrol acetate (MPA, 500 mg qd po)

SUMMARY:
Based on the above situation, the investigators propose the following scientific hypothesis: In young patients with early MMRd type EC, the use of immune checkpoint inhibitors combined with progesterone for fertility retention therapy can improve the therapeutic efficacy, reduce recurrence, and improve tumor prognosis.

Based on the above assumptions, this project intends to conduct a prospective exploratory clinical study in EC patients limited to the endometrial layer or superficial myometrium (FIGO 2023 IA1-IA2 stage). The subjects were treated with TQB2450 periodic intravenous drip + high-potency progesterone daily oral therapy. During the treatment period, hysteroscopy was performed every 12 weeks to evaluate the therapeutic efficacy. The primary endpoint was the 12-week CR rate; the secondary endpoints included the 24-week CR rate, the 36-week CR rate, the median CR time, the 1-year relapse rate, the 2-year relapse rate, the median relapse time, the pregnancy rate, the live birth rate, and drug-related adverse reactions. The exploratory indicators were the response of different MMRd tumors to immune checkpoint inhibitors and their possible mechanisms. The development of this study will provide a clinical basis for improving the fertility-preserving treatment regimen of MMRd EC.

DETAILED DESCRIPTION:
The incidence of endometrial cancer (EC) is on the rise and tends to be younger. With the release of China's multi-child policy and the delay of marriage and childbearing age in modern society, many endometrial cancer patients still have an urgent need to have children when they are found to be suffering from the disease. The standard treatment of EC is total hysterectomy, which makes women permanently lose their fertility. Therefore, the treatment of young EC patients with fertility preservation has become a new focus in the field of tumor reproduction. Conservative treatment based on large dose of progesterone is a classic treatment for early EC fertility preservation. For patients who meet the nursing standards, the complete response rate is 70-80%. This research group comprehensively evaluated the complete response rate of combined drug nursing treatment by hysteroscopy to reach 95%. However, it was also observed that about 1/3 of nurse-care patients had been treated for more than 9 months or continued to fail to achieve complete response (CR). Due to the prolonged duration of treatment, multiple hysteroscopic assessments during treatment increase the risk of endometrial injury, while long-term use of large doses of progesterone may lead to ovarian function suppression, all of which affect the success rate of pregnancy after complete remission. In addition, long-term oral large dose of progesterone can lead to increased risk of weight gain, liver function impairment, thrombosis, breast cancer, etc. Dizziness, headache and digestive tract symptoms during medication also affect patients' quality of life and reduce patients' treatment compliance. How to further optimize the early EC nursing treatment program, shorten the treatment time required to achieve complete remission, reduce adverse reactions, and improve the pregnancy rate after complete remission has become a new important topic facing EC nursing treatment.

The establishment of EC molecular typing provides a possibility for promoting EC precision therapy and improving patients' quality of life and prognosis. EC molecular typing has been proposed for more than 10 years, and endometrial cancer can be divided into four different types based on tumor molecular characteristics without any dependence on tumor morphological characteristics: POLE hypermutation (POLEmut), mismatch repair deficiency (MMRd), p53 abnormal, p53abn and no specific molecular profile (NSMP). Previous studies have confirmed high consistency between diagnostic endometrial specimens (biopsy or curettage) and whole uterine specimens. Molecular typing is helpful to predict the efficacy of endocrine therapy and has important reference value for judging whether patients of childbearing age can be treated with fertility preservation function.

MMRd type EC is relatively insensitive to progesterone therapy, and the selection of its treatment regimen is an important challenge for EC fertility-preserving therapy. MMRd type EC accounts for about 5% -16% of patients on fertility-preserving therapy. It has been reported that the remission rate of progesterone therapy in MMRd type EC and endometrial atypical hyperplasia patients is significantly lower than that in mismatch repair system intact type. In 2021, the first study on the effect of molecular typing on the prognosis of EC patients was published in South Korea. It was found that the overall progesterone response rate and the complete remission rate of disease at 6 months in MMRd type patients were significantly lower than those in p53 wild type patients. And even after complete remission, the recurrence rate of MMRd patients is higher. It is speculated that the reason may be that the tumor in this type of patients activates non-progesterone receptor-dependent molecular pathways, which in turn affects the focus's response to progesterone. For MMRd EC, it is necessary to explore new treatment options to improve the overall efficacy of EC care therapy.

Immune checkpoint inhibitors (ICIs) may be an effective treatment option to shorten the duration and improve the curative effect of MMRd-type EC. MMRd tumors have high tumor mutation burden caused by microsatellite instability (MSI-H) and are accompanied by a large number of tumor neoantigens and immune cell infiltration. Pathological features such as high tumor mutation burden and a large number of tumor neoantigens and immune cell infiltration provide feasibility for immunotherapy, among which programmed cell death receptor-1 (PD-1) and its ligand (PD-L1) inhibitors are one of the most popular targets of immunotherapy, and preliminary evidence confirms that they have clinical benefits for MMRd-type EC. In 2019, pembrolizumab was recommended by NCCN guidelines as an effective regimen for the systemic treatment of relapsed, metastatic, and high-risk EC in MSI-H/MMRd. Nivolumab, dostarlimab, and avelumab have also been confirmed to be effective in the treatment of EC, and are recommended in NCCN guidelines for second-line treatment in patients with relapsed and metastatic EC. The KEYNOTE-158 study enrolled 90 treated patients with advanced EC in MSI-H/dMMR and found an objective response rate of 48% (95% CI, 37% to 60%) to pabolizumab, with a median follow-up of 42.6 months (6.4-56 months), a median response time not reached (NR; range, 2.9-≥ 49.7 + months), a median progression-free survival time of 13.1 months (95% CI, 4.3-34 months), and a median overall survival time not reached; these results confirm that pabolizumab has effective and long-lasting antitumor activity, a favorable survival outcome, and controlled toxicity. In 2023, two high-quality randomized controlled clinical studies, NRG-GY018 and RUBY, both published results, confirming that the combination of anti-PD-1 inhibitors on the basis of platinum-containing chemotherapy can significantly improve the prognosis of locally advanced, metastatic or recurrent EC, especially in the dMMR population. After the publication of the two studies, pabolizumab and dotalizumab have been recommended by NCCN guidelines as the first-line systemic treatment regimen for advanced, metastatic or recurrent EC. ICIs have good anti-tumor effect in patients with advanced, metastatic or recurrent EC of MMRd type, but the efficacy in patients with MMRd type EC with retained fertility function still needs more research to confirm.

Case reports suggest that ICIs can be beneficial for fertility-preserving treatment of MMRd EC. Di Cao et al. reported a 36-year-old patient with Lynch syndrome, diagnosed with endometrioid carcinoma and colon cancer, who achieved complete tumor remission after treatment with sintilizumab, followed by successful pregnancy and live birth; no obvious adverse drug reactions were seen during the 11-month follow-up. Our research group has previously performed experimental ICI treatment on four patients with Lynch syndrome-related MMRd EC, and all four patients achieved complete remission. The treatment time was 18-42 weeks, and no tumor recurrence was seen during the follow-up period.

Benmelstobart (TQB2450) is a humanized monoclonal antibody that targets PD-L1, preventing PD-L1 from binding to the PD-1 and B7.1 receptors on the surface of T cells, restoring T cell activity, thereby enhancing the immune response, and has the potential to treat many types of tumors. Molecular formula: C6444H9968N1692O2002S46, molecular weight: 144,651 Da (non-glycosylation). There are currently 22 clinical studies registered, 6 of which are Phase III clinical trials.

Based on the above situation, we propose the following scientific hypothesis: In young patients with early MMRd type EC, the use of immune checkpoint inhibitors combined with progesterone for fertility retention therapy can improve the therapeutic efficacy, reduce recurrence, and improve tumor prognosis.

Based on the above assumptions, this project intends to conduct a prospective exploratory clinical study in EC patients limited to the endometrial layer or superficial myometrium (FIGO 2023 IA1-IA2 stage). The subjects were treated with TQB2450 periodic intravenous drip + high-potency progesterone daily oral therapy. During the treatment period, hysteroscopy was performed every 12 weeks to evaluate the therapeutic efficacy. The primary endpoint was the 12-week CR rate; the secondary endpoints included the 24-week CR rate, the 36-week CR rate, the median CR time, the 1-year relapse rate, the 2-year relapse rate, the median relapse time, the pregnancy rate, the live birth rate, and drug-related adverse reactions. The exploratory indicators were the response of different MMRd tumors to immune checkpoint inhibitors and their possible mechanisms. The development of this study will provide a clinical basis for improving the fertility-preserving treatment regimen of MMRd EC.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 45 years.
2. Pathological diagnosis of endometrioid carcinoma by biopsy, diagnostic curettage or hysteroscopy, non-invasive (G1-2); clinical diagnosis by G1-2); clinical diagnosis confirmed by at least two associate senior physicians;
3. Run possible, unknown EC;
4. Intense MRI, enhanced MMRI, enhanced MRI/CT, and pulmonary CT, or PET/CT assessments indicated that the lesions were limited to the endometrial layer or superficial myometrium, and there was no clear deep myometrium, cervix, or extrauterine involvement.
5. , WHFIGO 2023 IA1-IA2;
6. EC molecular typing, resulting in MMRd type (molecular typing is based on the World Health Organization (WHO) classification criteria for female genital tumors (5th edition) );
7. Those who require or insist on preserving reproductive function, or those who insist on preserving the uterus despite having no fertility requirements.

   informed
8. The hospital was followed up on schedule. 2. Exclusion criteria
9. and can be followed up regularly in this hospital.

Exclusion Criteria:

1. Endometrioid carcinoma FIGO grade G3, type II EC (including serous carcinoma, clear cell carcinoma, carcinosarcoma, undifferentiated carcinoma, dedifferentiated carcinoma, neuroendocrine carcinoma, etc.), or other non-epithelial uterine malignancies (adenosarcoma, stromal sarcoma, etc.);
2. Imaging evaluation indicates deep myometrial involvement, cervical involvement, or the possibility of extrauterine metastases.
3. History of important organ transplantation;
4. Uncontrolled diseases or active infections;
5. Concomitant with severe acute diseases such as stroke, myocardial infarction, etc.
6. Other malignant tumors of the reproductive system (except in patients with Lynch syndrome who also have ovarian cancer).
7. Those who require hysterectomy or other methods of treatment other than conservative medication.
8. Pregnant persons;
9. Those who have received conservative treatment (or medication maintenance treatment) with high-potency progesterone or oral contraceptives for more than 1 month due to endometrial hyperplasia in the past three months;
10. Smoking history, those who smoke more than 15 cigarettes per day;
11. Those who are contraindicated in the use of immunosuppressants or progesterone.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
3-month CR Rate | 12-16 weeks
  Complete response rate at 12-16 weeks of treatment

SECONDARY OUTCOMES:
6-month CR Rate | 24-28 weeks
  Complete response rate at 24-28 weeks of treatment
9-month CR Rate | 36-40 weeks
  Complete response rate at 36-40 weeks of treatment
median complete response duration | through study completion, an average of 2 years
1-year recurrence rate | 1 year after achieving CR
  recurrence rate at 1 year after achieving CR
2-year recurrence rate | 2 years after achieving CR
  recurrence rate at 2 years after achieving CR
median recurrence interval | through study completion, an average of 4 years
pregnancy rate | through study completion, an average of 4 years
live birth rate | through study completion, an average of 5 years
adverse event | through study completion, an average of 4 years
  drug-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yu Xue, M.D, Study Director — Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- Tenth People's Hospital of Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD is available upon reasonable request.